CLINICAL TRIAL: NCT02556112
Title: Effectiveness of a Group Lifestyle Balance Class in a Military Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Nicole Armitage, Chief, Clinical Investigations, David Grant U.S. Air Force Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FDG20150017H
Record Dates: First submitted 2015-09-15; First posted 2015-09-22 (Estimated); Results first posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Primary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group Lifestyle Balance (Active Comparator): Participants receive the Group Lifestyle Balance intervention as per the standard curriculum
  Interventions: Behavioral: Group Lifestyle Balance
- Better Body Better Life (Active Comparator): Participants receive the Better Body Better Life intervention as per the standard curriculum
  Interventions: Behavioral: Better Body Better Life
- Fitness Improvement Program (Active Comparator): Participants take the Fitness Improvement Program on-line
  Interventions: Behavioral: Fitness Improvement Program

INTERVENTIONS:
Behavioral: Group Lifestyle Balance — The content of the GLB program consists of educating participants about the association between high calorie and fat intake with excessive weight, how to determine the fat and calorie content of foods they eat, and how to make changes in their diet to reduce the fat and calorie content. Participants are also given information about increasing activity in their daily routines. In addition, they are given information about negative behaviors that lead to overeating and decreased activity and are taught ways to develop positive behaviors to facilitate weight loss and increased activity. GLB instructors function as lifestyle coaches for class participants. They provide individual feedback and encouragement on documented eating and activity habits. The instructors make themselves available to be contacted by participants outside of class to address participant concerns and issues as needed
  Other Names: GLB
  Arms: Group Lifestyle Balance
Behavioral: Better Body Better Life — The BBBL program is an Air Force weight management program.). It was created based on the Adult Learning Model and consists of 5 independent modules that are taught in-person to groups of up to 15-20 individuals. Each module is done in a classroom and is 2 hours long. One module per week is offered. Individuals can attend the modules in any order but they are required to complete a pre-survey and 3-day food record prior to attending their first class
  Other Names: BBBL
  Arms: Better Body Better Life
Behavioral: Fitness Improvement Program — The FIP is a standardized course that can be accessed on-line through the Advanced Distributed Learning Service (ADLS) and takes approximately 90 minutes to view all of the course material. The on-line FIP can be done all in one sitting or in segments. There is no restriction on the frequency with which the FIP is viewed however, because it is accessed through ADLS, it may be difficult to view at a non-military computer. The FIP consists of an introduction, three core components (nutrition, physical training, and spiritual well-being), and a summary. Each section has a short video presentation. The core components have short quizzes at the end to assess knowledge and the training asks participants to set goals. Participants are then responsible for using the information for their own self-directed program.
  Other Names: BE WELL
  Arms: Fitness Improvement Program

SUMMARY:
With this study researchers will evaluate the effects of the GLB intervention on weight loss, chronic disease indicators and self-perceived function and well-being in an active duty population. The purpose of this study is to examine the effectiveness of the GLB program [compared with two currently available programs, the Fitness Improvement Program (FIP) and the Better Body Better Life (BBBL) program], on the following health indicators: improvement of individual physical fitness as measured by change in abdominal circumference, weight and physical activity; decrease in risk associated with chronic disease as measured by changes in lipid and HbA1c levels; and improvement in self-perceived function and well-being as measured by the RAND 36 Item Short Form Health Survey (RAND SF- 36). In addition, the researchers seek to obtain feedback about the programs from the participants.

DETAILED DESCRIPTION:
Many active duty personnel struggle with weight gain and becoming overweight during the course of their active duty service. This can lead to difficulty in maintaining fitness standards and limit their ability to fully function in performing their mission. In addition, this may lead to increased risk for chronic disease development. Few published studies exist that evaluate interventions aimed at weight loss and chronic disease prevention in the active duty population. The Group Lifestyle Balance (GLB) program has been shown to be effective in facilitating weight loss and reducing chronic disease risk in civilian populations. However, the effectiveness of this class in preventing chronic illnesses, facilitating weight loss, increasing physical activity and promoting perceptions of improved functioning and well-being has not been studied in active duty populations. The purpose of this study will be to examine the effectiveness of the GLB program compared with the currently available Fitness Improvement Program (FIP) and Better Body Better Life (BBBL) on the following health indicators: individual physical fitness as measured by change in weight, abdominal circumference and minutes engaged in physical activity; changes in risk associated with chronic disease as measured by changes in lipid and HbA1c levels; and changes in self-perception of function and well-being as measured by the RAND SF-36 questionnaire.

This will be a quantitative randomized control intervention study to determine the effects of a GLB class on physical indicators of fitness, disease risk and overall perception of functional health and well-being in an active duty population, and to compare outcomes with the FIP intervention (care as usual) and newly implemented BBBL intervention currently offered to Airmen. This study will be conducted at David Grant Medical Center (DGMC), Travis AFB, California.

ELIGIBILITY:
Inclusion Criteria:

* • An active duty member of the USAF

  * Have at least one of the following conditions:

    * An abdominal circumference over 35 inches for men or 31.5 inches for women
    * BMI over 25 kg/m2
  * Are willing to commit to weekly 1 hour classes for 12 weeks and monthly 1 hour classes for an additional 3 months

Exclusion Criteria:

* • Women who are pregnant or breastfeeding

  * Participants who are within 8 months of a Permanent Change of Station or deployment
  * Anyone who has been restricted from participating in moderate activity equivalent to a brisk walk
  * Taking lipid-lowering or glucose-lowering medication
  * Anyone who for medical reasons cannot have a calorie-restricted diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Armitage NH, Kramer MK, Nelson MS, Hopkins D, Langeslay R, Thornton JA. Effectiveness of Lifestyle Interventions in an Active Duty Air Force Population. Am J Health Promot. 2021 Jul;35(6):784-793. doi: 10.1177/0890117121997308. Epub 2021 Mar 4. PMID 33657870

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began August 2015 and ended April 2018. Participants were recruited through flyers table tents in the Medical Group clinics and cafeteria and email blasts through unit fitness monitors.
Pre-assignment Details: Once participants were enrolled to the study, initial measurements (with the exception of lab work requiring blood draws) were taken before assignment to groups. The reason for this was to avoid bias on the part of the research team that might occur with knowledge of group assignment before obtaining initial data.
Groups:
- Group Lifestyle Balance: Participants receive the Group Lifestyle Balance intervention as per the standard curriculum
  Group Lifestyle Balance: Content consists of educating participants about the association between high calorie and fat intake with excessive weight, how to determine the fat and calorie content of foods they eat, and how to make changes in their diet to reduce the fat and calorie content. Participants are also given information about increasing activity in their daily routines. In addition, they are given information about negative behaviors that lead to overeating and decreased activity and are taught ways to develop positive behaviors to facilitate weight loss and increased activity. GLB instructors function as lifestyle coaches for class participants. They provide individual feedback and encouragement on documented eating and activity habits. The instructors make themselves available to be contacted by participants outside of class to address participant concerns
Period: Overall Study
Arm/Group | Group Lifestyle Balance | Better Body Better Life | Fitness Improvement Program
Started | 40 | 40 | 42
Completed | 30 | 23 | 30
Not Completed | 10 | 17 | 12

BASELINE CHARACTERISTICS:
Population: Baseline data was changed from all enrollees to study completers to be consistent with numbers of participants included in outcome measure analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Lifestyle Balance | Better Body Better Life | Fitness Improvement Program | Total
Number analyzed (Participants) | 30 | 23 | 30 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.30 (7.61) | 32.30 (5.05) | 32.90 (6.61) | 32.89 (6.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 9 | 13 | 40
  Male | 12 | 14 | 17 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 13 | 16 | 43
  African American | 9 | 5 | 5 | 19
  Hispanic/Latino | 5 | 3 | 4 | 12
  Asian | 1 | 2 | 3 | 6
  Multiple/Other | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 42 | 122
weight [Mean (Standard Deviation); unit: pounds] | 190.95 (31.20) | 200.29 (32.26) | 204.46 (36.68) | 199.66 (33.72)
abdominal circumference [Mean (Standard Deviation); unit: inches] | 35.51 (3.63) | 36.49 (4.17) | 36.86 (4.02) | 36.30 (3.96)
lipid [Mean (Full Range); unit: mg/dL]
  Total Cholesterol | 187.5 [134 to 286] | 180.00 [138 to 293] | 176 [107 to 255] | 181.27 [107 to 286]
  HDL | 51 [27 to 96] | 54 [36 to 121] | 52 [35 to 88] | 52.19 [27 to 121]
  LDL | 111.8 [68.8 to 189] | 100 [60 to 205] | 92 [36 to 181] | 101.37 [36 to 205]
  Triglycerides | 92.5 [39 to 280] | 89 [47 to 290] | 84 [30 to 226] | 88.46 [30 to 290]
hgbA1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 5.33 (.36) | 5.28 (.24) | 5.24 (.47) | 5.28 (.36)

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: measured on a calibrated human weight scale
Time Frame: 6 months
Population: Weight measurement in pounds at 6 months
Measure: Mean (Standard Error); unit: pounds
Arm/Group | Group Lifestyle Balance | Better Body Better Life | Fitness Improvement Program
Number analyzed (Participants) | 30 | 23 | 30
pounds | 191.47 (5.39) | 198.08 (7.27) | 204.08 (7.24)

2. Primary Outcome: Abdominal Circumference
Description: measurement taken as per Air Force Instruction for the Fitness Assessment
Time Frame: measured at 6 months
Population: Abdominal circumference in inches at 6 months
Measure: Mean (Standard Error); unit: inches
Arm/Group | Group Lifestyle Balance | Better Body Better Life | Fitness Improvement Program
Number analyzed (Participants) | 30 | 30 | 23
inches | 34.96 (.70) | 35.68 (.86) | 36.09 (.80)

3. Secondary Outcome: Well-being
Description: as measured by the Rand SF 36 questionnaire. Scores range from 0-100 with higher scores indicating greater well-being or function.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Group Lifestyle Balance: Participants receive the Group Lifestyle Balance intervention as per the standard curriculum
  Group Lifestyle Balance: The content of the GLB program consists of educating participants about the association between high calorie and fat intake with excessive weight, how to determine the fat and calorie content of foods they eat, and how to make changes in their diet to reduce the fat and calorie content. Participants are also given information about increasing activity in their daily routines. In addition, they are given information about negative behaviors that lead to overeating and decreased activity and are taught ways to develop positive behaviors to facilitate weight loss and increased activity. GLB instructors function as lifestyle coaches for class participants. They provide individual feedback and encouragement on documented eating and activity habits.
Arm/Group | Group Lifestyle Balance | Better Body Better Life | Fitness Improvement Program
Number analyzed (Participants) | 30 | 23 | 30
score on a scale | 77 (7.68) | 82 (6.78) | 76 (7.75)

4. Secondary Outcome: Lipids
Description: serum levels obtained through venipuncture
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: total cholesterol mg/dL
Arm/Group | Group Lifestyle Balance | Better Body Better Life | Fitness Improvement Program
Number analyzed (Participants) | 30 | 23 | 30
total cholesterol mg/dL | 188.17 (34.59) | 180.52 (36.15) | 170.67 (31.73)

5. Secondary Outcome: Physical Activity
Description: As measured by minutes per week of physical activity
Time Frame: 6 months
Measure: Median (Standard Error); unit: minutes per week
Arm/Group | Group Lifestyle Balance | Better Body Better Life | Fitness Improvement Program
Number analyzed (Participants) | 30 | 23 | 30
minutes per week | 45 (7.68) | 50 (6.78) | 45 (7.75)

6. Secondary Outcome: HbA1C
Description: serum levels obtained through venipuncture
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Group Lifestyle Balance | Better Body Better Life | Fitness Improvement Program
Number analyzed (Participants) | 30 | 23 | 30
percentage of glycosylated hemoglobin | 5.26 (.43) | 5.22 (.45) | 5.26 (.40)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for approximately 6 months for each participant. Data were collected from the time participants started the study until they completed data collection at the 6 month time frame.
Arm/Group | Group Lifestyle Balance | Better Body Better Life | Fitness Improvement Program
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Protocol and statistical analysis plan (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT02556112/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT02556112/ICF_001.pdf